CLINICAL TRIAL: NCT02646618
Title: Get Social: Randomized Trial of a Social Network Delivered Lifestyle Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Connecticut (Other)
Collaborators: Worcester Polytechnic Institute (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Sherry Pagoto, Professor, University of Connecticut
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H17-210; 1R01DK103944-01A1 (NIH)
Record Dates: First submitted 2016-01-04; First posted 2016-01-05 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Get Social (Active Comparator): Get Social participants will receive a weight loss intervention in a "protected" Twitter group. The intervention content will be structured to deliver in an online context. The online coaches will post daily content, respond to questions, address concerns, and encourage engagement. The weight loss intervention is based on the Diabetes Prevention Program (DPP), an evidence-based weight loss program focused on lifestyle changes. The goals for the intervention are 175 minutes of moderate physical activity per week and an overall weight loss of 7%. Each participant will get an individualized calorie goal that would facilitate a 1-2 lbs. weight loss weekly. Participants will also be encouraged to use an app such as MyFitnessPal to track daily diet.
  Interventions: Behavioral: Get Social; Device: Smartphone
- Traditional (Active Comparator): Participants will attend weight loss groups weekly for 8 weeks, then biweekly for 16 weeks, then monthly between months 6 and 12. The weight loss intervention is based on the Diabetes Prevention Program (DPP), an evidence-based weight loss program focused on lifestyle changes. The goals for the intervention are 175 minutes of moderate physical activity per week and an overall weight loss of 7%. Each participant will get an individualized calorie goal that would facilitate a 1-2 lbs. weight loss weekly. Participants will also be encouraged to use an app such as MyFitnessPal to track daily diet.
  Interventions: Behavioral: Traditional; Device: Smartphone

INTERVENTIONS:
Behavioral: Get Social — Online-delivered weight loss intervention
  Arms: Get Social
Behavioral: Traditional — Group-delivered weight loss intervention
  Arms: Traditional
Device: Smartphone — A smartphone is needed to use MyFitnessPal for all participants and to access Twitter for the Get Social participants

SUMMARY:
The present study is a non-inferiority trial comparing the efficacy of a lifestyle intervention delivered entirely via an online social network to a traditional lifestyle intervention delivered via group meetings.

DETAILED DESCRIPTION:
Lifestyle interventions have had established efficacy for over a decade but are still not widely disseminated, largely due to high cost and patient and provider burden. Online social networks are an alternative way to deliver lifestyle counseling and delivery via this modality may virtually eliminate patient visits, the main source of cost and burden in traditional modalities. Interactions in online social networks are frequent, brief, and asynchronous because users login to their online communities during downtime during work and leisure time, or when they simply feel a need for social connection. As such, social media becomes embedded into people's daily lives. This provides an opportunity to embed health behavior change programming into people's daily lives. Thus far in the literature, existing online social networks have been used as component of web- or mobile app-based lifestyle interventions but not as the primary modality for intervention delivery. The purpose of this work is to conduct a non-inferiority trial to compare a lifestyle intervention delivered entirely via private groups on the online social network Twitter to a traditional in-person group-based lifestyle intervention. Using a randomized trial (N=328), investigators will test whether a lifestyle intervention delivered via an online social network (Get Social condition) will result in a mean percent weight loss at 12 months that is not appreciably worse than the gold-standard in-person group-based lifestyle intervention (Traditional condition), i.e., the social network arm will not lose on average 2% less than the in-person arm. Secondary non-inferiority outcomes include weight loss at 12 months, and dietary intake and physical activity at 12-months. Investigators hypothesize that the Get Social condition will be less expensive than the Traditional condition. To understand for whom an online social network modality is most suited, investigators will test predictors of weight loss in the Get Social condition including engagement, age, sociability, neuroticism, openness, and smartphone and social network use. Investigators hypothesize that people who are younger, more sociable, engage more on the social network, higher in neuroticism/openness, and heavier overall smartphone and social network users will lose more weight in the Get Social condition. Findings from this study may support an intervention delivery modality that is more conducive to settings like worksites, health plans, and clinics that serve large populations but have limited space, staffing, and resources for traditional in person interventions.

ELIGIBILITY:
Inclusion:

1. Smartphone users
2. Ages 18-65
3. Body Mass Index (BMI) 27-45
4. Must currently log into a social media platform on a daily basis basis and engage (like, reply, post) at least 4 days per week.

Participants will be excluded if they:

1. Do not have a smartphone;
2. Are unable to get medical clearance from their Primary Care Physician (PCP);
3. Have plans to move during study;
4. Are not interested in losing weight;
5. Have Type 1 or uncontrolled 2 Diabetes (as determined by PCP);
6. Have medical conditions that would prevent increasing physical activity or making dietary changes;
7. Are pregnant/lactating or plans to become pregnant during study;
8. Are currently taking medication affecting weight;
9. Currently participating in a weight loss program or using an online social network to assist them with weight loss (e.g. Weight Watchers, Sparkpeople, etc);
10. Unable to walk at least ¼ mile unaided without stopping;
11. Experienced a weight loss of 5% or more in past 3 month;
12. A history of/or plans on having bariatric surgery;
13. Did not complete the baseline measures;
14. Not willing to use Twitter, or if a current Twitter user, not willing to create a new account specifically for study purposes;
15. Participated in another weight loss study under the direction of the PI of this study;
16. Current smoker (smokes 3 or more cigarettes per day);
17. Unavailable to attend weekly group meetings;
18. Prefers one condition over another;
19. Score of 30 or higher on the Beck Depression Inventory (BDI) or endorsement of 2 or 3 on BDI #9 indicating suicidal thoughts;
20. Presence of binge eating disorder
21. Did not complete the orientation webinar;
22. Are unable to provide consent due to mental illness or a cognitive impairment;
23. Does not speak English; or
24. Are a prisoner.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sherry Pagoto, Principal Investigator — University of Connecticut
Locations (1):
- University of Connecticut, Storrs, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pagoto SL, Goetz JM, Xu R, Wang ML, Palmer L, Lemon SC. Randomized non-inferiority trial comparing an asynchronous remotely-delivered versus clinic-delivered lifestyle intervention. Int J Obes (Lond). 2025 Jan;49(1):76-83. doi: 10.1038/s41366-024-01617-0. Epub 2024 Aug 27. PMID 39191926
- [Derived] Jake-Schoffman DE, Brown SD, Baiocchi M, Bibeau JL, Daubenmier J, Ferrara A, Galarce MN, Hartogensis W, Hecht FM, Hedderson MM, Moran PJ, Pagoto SL, Tsai AL, Waring ME, Kiernan M. Methods-Motivational Interviewing Approach for Enhanced Retention and Attendance. Am J Prev Med. 2021 Oct;61(4):606-617. doi: 10.1016/j.amepre.2021.04.005. PMID 34544560
- [Derived] Wang ML, Waring ME, Jake-Schoffman DE, Oleski JL, Michaels Z, Goetz JM, Lemon SC, Ma Y, Pagoto SL. Clinic Versus Online Social Network-Delivered Lifestyle Interventions: Protocol for the Get Social Noninferiority Randomized Controlled Trial. JMIR Res Protoc. 2017 Dec 11;6(12):e243. doi: 10.2196/resprot.8068. PMID 29229591

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Get Social | Traditional
Started | 167 | 162
6 Month Follow-up | 152 | 150
Completed | 157 | 148
Not Completed | 10 | 14
Not completed — Lost to Follow-up | 10 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Get Social | Traditional | Total
Number analyzed (Participants) | 167 | 162 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.3 (11.2) | 45.5 (11.6) | 45.4 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 132 | 268
  Male | 31 | 30 | 61
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 16
  Not Hispanic or Latino | 158 | 154 | 312
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 4 | 3 | 7
  White | 152 | 150 | 302
  More than one race | 3 | 5 | 8
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 167 | 162 | 329
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 34.9 (4.8) | 35.1 (4.4) | 35.0 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: A digital scale (Scaletronix, Model-5002) will be used to record weight
Time Frame: Baseline
Population: Randomized participants
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
lbs | 214.7 (36.9) | 215.4 (35.8)

2. Primary Outcome: Percent Weight Change
Description: A digital scale (Scaletronix, Model-5002) will be used to record weight
Time Frame: Baseline to 6-months
Population: Randomized participants
Measure: Mean (Standard Error); unit: Percent change in weight
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Percent change in weight | -2.6 (0.5) | -4.5 (0.5)
Statistical Analysis 1: Comparison: Get Social vs Traditional; Test type: Non-Inferiority — We set δ=2% as a relative margin to the 5% weight loss as clinically meaningful cut point and because 2% is not so small a difference in average weight loss between study conditions that we would have to recruit a prohibitively large sample; p = 0.0038, Mixed Models Analysis; Mean Difference (Net) = 2.0, 95% CI 2-sided [0.6 to 3.3]

3. Primary Outcome: Percent Weight Change
Description: A digital scale (Scaletronix, Model-5002) will be used to record weight
Time Frame: Baseline to 12-months
Population: Randomized participants
Measure: Mean (Standard Error); unit: Percent change in weight
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Percent change in weight | -2.6 (0.6) | -3.7 (0.6)
Statistical Analysis 1: Comparison: Get Social vs Traditional; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p = 0.1485, Mixed Models Analysis; Mean Difference (Net) = 1.2, 95% CI 2-sided [-0.4 to 2.8]

4. Secondary Outcome: Cost Associated With Intervention
Description: Total time to deliver the intervention and administrative time was tracked during the study for each condition and cost was calculated using national median salary for dietitians & nutritionists and administrative assistants & secretaries, and national fringe data for all civilian workers across all industries from Bureau of Labor Statistics. Hourly rate based on salary plus fringe divided by 2080 hours (40 hours/week x 52 weeks). Administrative tasks charged at administrative assistant salary rate, all other treatment delivery tasks charged at dietitian rate. Dollars per participant was calculated by dividing total cost for each condition by the number of participants in that condition.
Time Frame: 12-months
Population: Randomized participants
Measure: Number; unit: dollars per participant
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
dollars per participant | 114 | 165

5. Secondary Outcome: Time Spent During Intervention
Description: Administrative and intervention-delivery was measured. Amount of administrative and intervention delivery time per participant was calculated.
Time Frame: 12-months
Population: Randomized participants
Measure: Mean (Standard Deviation); unit: Hours per participant
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Hours per participant | 3.0 (1.1) | 3.9 (1.8)
Statistical Analysis 1: Comparison: Get Social vs Traditional; Test type: Superiority; p = 0.2480, t-test, 2 sided

6. Secondary Outcome: Retention at Follow-up
Description: Retention will be calculated as the percentage of participants who complete the final weigh-in in each condition.
Time Frame: 12-months
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Participants | 157 | 148

7. Secondary Outcome: Acceptability of the Intervention
Description: Acceptability and their satisfaction with intervention was measured by asking participants "If given the opportunity to continue participating in the program, how willing would you be to continue?" Response options were from 1 ("Definitely would") to 5 ("Definitely would not"). The outcome is the number of positive responses which include responses of 1 or 2 ("Probably would") on this measure.
Time Frame: 6-months
Population: Randomized participants who completed the acceptability question
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 127 | 140
Participants | 100 | 104

8. Secondary Outcome: Burden of Intervention
Description: Burden was measured through the question "Participating in the program was time consuming." Response options were 1 ("Strongly agree") to 5 ("Strongly disagree"). We are reporting number of participants who agreed with the statement by responding with a 1 ("Strongly agree") or 2 ("Agree")
Time Frame: 6-months
Population: Randomized participants who completed the burden question
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 127 | 140
Participants | 37 | 62

9. Secondary Outcome: Dietary Intake
Description: National Cancer Institute's (NCI) automated self-administered 24-hour dietary recall (ASA24™) was used to measure caloric intake.
Time Frame: Baseline
Population: Randomized participants with valid recall data
Measure: Mean (Standard Deviation); unit: kcal
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 161
kcal | 2168 (642) | 2042 (548)

10. Secondary Outcome: Change in Dietary Intake
Description: National Cancer Institute's (NCI) automated self-administered 24-hour dietary recall (ASA24™) measured caloric intake. Difference in caloric intake during baseline and 6 month evaluations was calculated.
Time Frame: Baseline to 6-months
Population: Randomized participants with valid recall data
Measure: Mean (Standard Error); unit: kcal
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
kcal | -316 (52) | -410 (51)
Statistical Analysis 1: Comparison: Get Social vs Traditional; Test type: Non-Inferiority — For secondary noninferiority outcomes, we used 90% power to calculate noninferiority margins given N=131 per arm, setting alpha=.05 and using observed SDs from the literature. For change in energy (kcal/day) intake, the study is powered at 90% to detect whether the Get Social condition is not inferior to the Traditional condition with a noninferiority margin of 182 kcal/day (SD=500 kcal/day); p = 0.2025, Mixed Models Analysis; Mean Difference (Net) = 93, 95% CI 2-sided [-50 to 237]

11. Secondary Outcome: Change in Dietary Intake
Description: National Cancer Institute's (NCI) automated self-administered 24-hour dietary recall (ASA24™) will record dietary intake. Change in caloric intake between baseline and 12 months was calculated.
Time Frame: Baseline to 12-months
Population: Randomized participants with valid recall data
Measure: Mean (Standard Error); unit: kcal
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
kcal | -396 (55) | -321 (54)
Statistical Analysis 1: Comparison: Get Social vs Traditional; Test type: Non-Inferiority — [test comment as in outcome 10, analysis 1]; p = 0.3323, Mixed Models Analysis; Mean Difference (Net) = -75, 95% CI 2-sided [-226 to 77]

12. Secondary Outcome: Physical Activity
Description: Arizona Physical Activity Questionnaire will be used to provide estimates of total energy expenditure to calculate number of participants reaching the guideline of 150 minutes per week of moderate to vigorous physical activity.
Time Frame: Baseline
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Participants | 81 | 70

13. Secondary Outcome: Physical Activity
Description: as for outcome 12
Time Frame: Baseline to 6-months
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Participants | 88 | 93
Statistical Analysis 1: Comparison: Get Social vs Traditional; We examined the proportion of participants engaging in 150+ minutes/week of moderate/vigorous intensity physical activity (MVPA) using generalized estimating equations with a logit link function and incorporating repeated measures over time. For participants missing MVPA at either follow-up timepoint, we used a baseline observation carried forward approach to impute their activity level (150+ vs <150 MVPA mins/week) at that timepoint; Test type: Non-Inferiority — For secondary noninferiority outcomes, we used 90% power to calculate noninferiority margins given N=131 per arm, setting alpha=.05 and using observed SDs from the literature. For change in moderate to vigorous intensity physical activity minutes per day at 12 months, the noninferiority margin is 9.2 min/day(SD=25 min/day). However, we could not analyze the data in that manner and used the test described above; p = 0.3905, Generalized estimating equation

14. Secondary Outcome: Physical Activity
Description: as for outcome 12
Time Frame: Baseline to 12-months
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Participants | 87 | 78
Statistical Analysis 1: Comparison: Get Social vs Traditional; [analysis description as in outcome 13, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 13, analysis 1]; p = 0.4741, Generalized estimating equation

15. Secondary Outcome: Intervention Engagement
Description: Engagement will be measured by tracking group attendance and quantifying communication in the online group throughout the intervention in terms of percent of intervention modules participated in.
Time Frame: 6-months
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: Percentage of modules participated in
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Percentage of modules participated in | 93.8 [62.5 to 100.0] | 68.8 [37.5 to 81.3]

16. Secondary Outcome: Intervention Engagement
Description: as for outcome 15
Time Frame: 12-months
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: Percentage of modules participated in
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Percentage of modules participated in | 81.8 [50.0 to 100.0] | 63.6 [27.3 to 81.8]

17. Secondary Outcome: Social Support for Weight Loss
Description: Weight Management Support Inventory to assess social support for weight management. The directions ask respondents to rate on a 5-point scale how frequently they experienced a certain interaction with other people in the past 4 weeks, ranging from 1 (never) to 5 (daily). The items also ask how helpful that event was when it occurred, rated on a 5-point scale ranging from 1 (not helpful) to 5 (extremely helpful). Higher scores indicate more frequent or more helpful social support events. We asked this about four potential social groups: family, friends, friends on Twitter, and friends on Facebook.
Time Frame: Baseline
Population: Randomized participants who completed each of the WMSI subscales.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
score on a scale
  Family - Frequency | 1.5 [1.2 to 1.8] | 1.4 [1.2 to 1.7]
  Family - Helpfulness: number analyzed (Participants) | 159 | 154
  Family - Helpfulness | 2.1 [1.5 to 3.0] | 2.0 [1.4 to 2.7]
  Friends - Frequency | 1.3 [1.0 to 1.6] | 1.2 [1.0 to 1.6]
  Friends - Helpfulness: number analyzed (Participants) | 145 | 143
  Friends - Helpfulness | 1.9 [1.3 to 2.9] | 2.0 [1.2 to 3.0]
  Twitter Friends - Frequency: number analyzed (Participants) | 102 | 91
  Twitter Friends - Frequency | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Twitter Friends - Helpfulness: number analyzed (Participants) | 53 | 43
  Twitter Friends - Helpfulness | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.0]
  Facebook Friends - Frequency: number analyzed (Participants) | 167 | 159
  Facebook Friends - Frequency | 1.0 [1.0 to 1.2] | 1.0 [1.0 to 1.2]
  Facebook Friends - Helpfulness: number analyzed (Participants) | 113 | 110
  Facebook Friends - Helpfulness | 1.2 [1.0 to 2.3] | 1.3 [1.0 to 2.0]

18. Secondary Outcome: Social Support for Weight Loss
Description: as for outcome 17
Time Frame: 6-months
Population: Randomized participants who completed the relevant WMSI scales
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 127 | 141
score on a scale
  Family - Frequency | 1.5 [1.2 to 1.8] | 1.5 [1.2 to 1.8]
  Family - Helpfulness: number analyzed (Participants) | 120 | 127
  Family - Helpfulness | 2.8 [2.0 to 3.4] | 2.7 [2.0 to 3.4]
  Friends - Frequency: number analyzed (Participants) | 126 | 141
  Friends - Frequency | 1.4 [1.1 to 1.6] | 1.2 [1.0 to 1.6]
  Friends - Helpfulness: number analyzed (Participants) | 108 | 111
  Friends - Helpfulness | 2.8 [2.0 to 3.6] | 3.0 [2.0 to 3.7]
  Twitter Friends - Frequency: number analyzed (Participants) | 117 | 75
  Twitter Friends - Frequency | 1.6 [1.2 to 2.0] | 1.0 [1.0 to 1.0]
  Twitter Friends - Helpfulness: number analyzed (Participants) | 96 | 13
  Twitter Friends - Helpfulness | 2.8 [2.1 to 3.7] | 1.0 [1.0 to 1.0]
  Facebook Friends - Frequency: number analyzed (Participants) | 123 | 135
  Facebook Friends - Frequency | 1.0 [1.0 to 1.2] | 1.0 [1.0 to 1.1]
  Facebook Friends - Helpfulness: number analyzed (Participants) | 56 | 57
  Facebook Friends - Helpfulness | 2.1 [1.1 to 3.3] | 2.7 [1.1 to 3.3]

19. Secondary Outcome: Social Support for Weight Loss
Description: as for outcome 17
Time Frame: 12-months
Population: Randomized participants who complete the relevant module of the WMSI
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 113 | 126
units on a scale
  Family - Frequency | 1.4 [1.2 to 1.7] | 1.3 [1.1 to 1.6]
  Family - Helpfulness: number analyzed (Participants) | 104 | 112
  Family - Helpfulness | 3.0 [2.0 to 3.8] | 3.0 [2.1 to 3.5]
  Friends - Frequency | 1.2 [1.0 to 1.6] | 1.2 [1.0 to 1.4]
  Friends - Helpfulness: number analyzed (Participants) | 88 | 90
  Friends - Helpfulness | 3.1 [2.0 to 4.0] | 3.0 [2.0 to 3.5]
  Twitter Friends - Frequency: number analyzed (Participants) | 96 | 113
  Twitter Friends - Frequency | 1.0 [1.0 to 1.4] | 1.0 [1.0 to 1.0]
  Twitter Friends - Helpfulness: number analyzed (Participants) | 3 | 26
  Twitter Friends - Helpfulness | 2.8 [2.0 to 4.0] | 1.0 [1.0 to 3.0]
  Facebook Friends - Frequency: number analyzed (Participants) | 113 | 117
  Facebook Friends - Frequency | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.1]
  Facebook Friends - Helpfulness: number analyzed (Participants) | 26 | 38
  Facebook Friends - Helpfulness | 3.0 [2.0 to 4.0] | 3.0 [2.0 to 3.5]

20. Secondary Outcome: Neuroticism/Emotional Stability and Openness to Experience
Description: Openness to Experience and Neuroticism/Emotional Stability were measured using the Ten-Item Personality Inventory. The Ten-Item Personality Inventory consists of 10 items that measure the five dimensions of the Five Factor model of personality. Participants are asked to respond to a series of words with personality descriptions with the prompt "I see myself as" with response options of 1 ("Disagree Strongly") to 7 ("Agree Strongly"). Opposite items are reverse coded. Items for Emotional Stability/Neuroticism are "anxious, easily upset" and "calm, emotionally stable". Items for Openness to experience are "open to new experiences, complex" or "conventional, uncreative." The average of the scores represents each dimension with higher scores indicating higher levels of Openness or Emotional Stability (and lower levels of Neuroticism).
Time Frame: Baseline
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
score on a scale
  Emotional Stability/Neuroticism | 5 [4.5 to 6] | 5 [4 to 6]
  Openness to Experience | 5.5 [5 to 6] | 6 [5 to 6.5]

21. Secondary Outcome: Social Media Use
Description: Twitter use was measured by asking participants which social networks they had an account on
Time Frame: Baseline
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Participants | 102 | 91

22. Secondary Outcome: Social Media Use
Description: Participants were asked which social networks they had an account on and number with a Twitter account was reported.
Time Frame: 6-months
Population: Randomized participants who completed questions about social media use
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 130 | 143
Participants | 117 | 75

23. Secondary Outcome: Social Media Use
Description: Participants were asked which social networks they had an account on and number with a Twitter account was reported.
Time Frame: 12-months
Population: Randomized participants who completed questions regarding social media use
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 118 | 129
Participants | 100 | 68

24. Secondary Outcome: Blood Pressure
Description: The average of two blood pressure readings was used as the measure of blood pressure. If participants only had one blood pressure reading that was used as the measure of blood pressure.
Time Frame: Baseline
Population: Randomized participants
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
mmHg
  Systolic blood pressure | 134.4 (13.0) | 133.1 (12.9)
  Diastolic blood pressure | 82.4 (8.3) | 82.3 (10.3)

25. Secondary Outcome: Blood Pressure
Description: as for outcome 24
Time Frame: 6-months
Population: Randomized participants who were able to complete blood pressure measurement
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 136 | 142
mmHg
  Systolic blood pressure | 130.6 (12.7) | 130.2 (13.6)
  Diastolic blood pressure | 80.1 (8.8) | 81.1 (9.2)

26. Secondary Outcome: Blood Pressure
Description: as for outcome 24
Time Frame: 12-months
Population: Randomized participants who were able to have their blood pressure measured
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 128 | 133
mmHg
  Systolic blood pressure | 130.6 (14.0) | 129.7 (13.7)
  Diastolic blood pressure | 80.3 (9.3) | 81.1 (9.6)

27. Secondary Outcome: STOP (Snoring, Tired, Observed Apnea, Pressure) Questionnaire
Description: Participants completed the four item STOP sleep apnea questionnaire. Participants who answered yes to 0-1 items were classified as low risk for sleep apnea. Participants who answered yes to 2-4 items were classified as high risk for sleep apnea.
Time Frame: Baseline
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Participants
  Low risk for sleep apnea | 116 | 105
  High risk for sleep apnea | 51 | 57

28. Secondary Outcome: STOP (Snoring, Tired, Observed Apnea, Pressure) Questionnaire
Description: as for outcome 27
Time Frame: 6-month
Population: Randomized participants who completed the STOP questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 128 | 141
Participants
  Low risk of sleep apnea | 94 | 101
  High risk of sleep apnea | 34 | 40

29. Secondary Outcome: STOP (Snoring, Tired, Observed Apnea, Pressure) Questionnaire
Description: as for outcome 27
Time Frame: 12-month
Population: Randomized participants who completed the STOP questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 117 | 129
Participants
  Low risk of sleep apnea | 83 | 96
  High risk of sleep apnea | 34 | 33

30. Secondary Outcome: Insomnia Severity Index
Description: To measure sleep quality, participants completed the Insomnia Severity Index. Higher scores (maximum 28) represent increased levels of insomnia, from 0-7 ("Absence of insomnia"), through 8-14 ("Sub-threshold insomnia"), 15-21 ("Moderate insomnia"), and 22-28 ("Severe insomnia").
Time Frame: Baseline
Population: Randomized participants
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
score on a scale | 5 [2 to 9] | 6 [3 to 9]

31. Secondary Outcome: Insomnia Severity Index
Description: as for outcome 30
Time Frame: 6-months
Population: Randomized participants who completed the ISI at 6 months.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 128 | 141
score on a scale | 5 [2 to 10] | 6 [3 to 10]

32. Secondary Outcome: Insomnia Severity Index
Description: as for outcome 30
Time Frame: 12-months
Population: Randomized participants who completed the ISI at 12 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 117 | 129
score on a scale | 5 [2 to 9] | 5 [3 to 10]

33. Secondary Outcome: Sleep Duration
Description: To measure sleep quality we used select questions from the Pittsburgh Sleep Quality Index which allowed the calculation of sleep duration.
Time Frame: Baseline
Population: Randomized participants who completed the PSQI items
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 161
hours | 7.0 [6.0 to 7.0] | 7.0 [6.0 to 7.0]

34. Secondary Outcome: Sleep Duration
Description: as for outcome 33
Time Frame: 6-months
Population: Randomized participants who completed the PSQI items
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 128 | 140
hours | 6.5 [6.0 to 7.0] | 7.0 [6.0 to 7.5]

35. Secondary Outcome: Sleep Duration
Description: as for outcome 33
Time Frame: 12-months
Population: Randomized participants who completed the PSQI items
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 116 | 128
hours | 7.0 [6.0 to 7.0] | 7.0 [6.0 to 7.0]

36. Secondary Outcome: History of Sleep Apnea
Description: Participants were asked whether they had ever been diagnosed with sleep apnea with response options Yes or No.
Time Frame: Baseline
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Participants
  No | 143 | 144
  Yes | 24 | 18

37. Secondary Outcome: Previous or Current Treatment for Sleep Apnea
Description: Participants were asked 1. Are you being treated for sleep apnea presently? (Yes/No) and 2. Have you ever received treatment for sleep apnea?
Time Frame: Baseline
Population: Randomized participants (For current treatment, only randomized participants who reported previous sleep apnea diagnosis)
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Participants
  Current Treatment of Sleep Apnea (Participants with sleep apnea diagnosis): number analyzed (Participants) | 24 | 18
  Current Treatment of Sleep Apnea (Participants with sleep apnea diagnosis): No | 5 | 7
  Current Treatment of Sleep Apnea (Participants with sleep apnea diagnosis): Yes | 19 | 11
  Past Treatment of Sleep Apnea: No | 145 | 146
  Past Treatment of Sleep Apnea: Yes | 22 | 16

38. Secondary Outcome: Diagnosis or Current Treatment for Sleep Apnea
Description: Participants were asked: Have you ever been diagnosed with sleep apnea? If they answered yes, they were asked if they were currently being treated for sleep apnea.
Time Frame: 6-months
Population: Randomized participants who completed questions relating to sleep apnea at 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 128 | 141
Participants
  Diagnosis of sleep apnea: No | 103 | 124
  Diagnosis of sleep apnea: Yes | 25 | 17
  Current treatment for sleep apnea: number analyzed (Participants) | 25 | 17
  Current treatment for sleep apnea: No | 9 | 8
  Current treatment for sleep apnea: Yes | 16 | 9

39. Secondary Outcome: Diagnosis or Current Treatment for Sleep Apnea
Description: as for outcome 38
Time Frame: 12-months
Population: Randomized participants who completed the questions about sleep apnea
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 117 | 129
Participants
  Diagnosis of sleep apnea: No | 94 | 114
  Diagnosis of sleep apnea: Yes | 23 | 15
  Current treatment of sleep apnea: number analyzed (Participants) | 23 | 15
  Current treatment of sleep apnea: No | 8 | 6
  Current treatment of sleep apnea: Yes | 15 | 9

40. Secondary Outcome: Beck Depression Inventory
Description: To measure depressive symptoms, participants completed the Beck Depression Inventory. Total scores can be interpreted as 1-10 ("normal ups and downs"), 11-16 ("Mild mood disturbance"), 17-20 ("Borderline clinical depression"), 21-30 ("Moderate depression"), 31-40 ("Severe depression"), 41+ ("Extreme depression").
Time Frame: Baseline
Population: Randomized participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
score on a scale | 6.1 (5.3) | 7.7 (7.3)

41. Secondary Outcome: Beck Depression Inventory
Description: as for outcome 40
Time Frame: 6-months
Population: Randomized participants who completed the BDI
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 128 | 141
score on a scale | 5.6 (5.8) | 6.3 (7.5)

42. Secondary Outcome: Beck Depression Inventory
Description: as for outcome 40
Time Frame: 12-months
Population: Randomized participants who completed the BDI
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 117 | 129
score on a scale | 4.8 (5.3) | 5.7 (5.9)

43. Secondary Outcome: Weight-Loss Related Social Media Use
Description: Participants were asked "Have you ever posted about or had discussions about your weight loss or desire to lose weight?" Number who answered yes are reported.
Time Frame: Baseline
Population: Randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Participants | 58 | 59

44. Secondary Outcome: Weight-Loss Related Social Media Use
Description: as for outcome 43
Time Frame: 6-months
Population: Randomized participants who responded to the question about weight-loss related social media use
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 126 | 139
Participants | 78 | 36

45. Secondary Outcome: Weight-Loss Related Social Media Use
Description: as for outcome 43
Time Frame: 12-months
Population: Randomized participants who answered the question about weight-loss related social media use.
Measure: Count of Participants; unit: Participants
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 114 | 125
Participants | 48 | 28

46. Secondary Outcome: Treatment Fidelity
Description: The intervention was divided into different content units delivered either during a meeting (Traditional Condition) or a series of tweets (Get Social Condition). For the Get Social Condition, tweets with intervention content were produced to meet all objectives for each content unit and programmed to go out at set times for each group so 100% of the objectives for each content unit were met. For the Traditional Condition, checklists were created with objectives for each content unit and staff listened to 2 to 3 randomly selected group recordings for each study wave to determine if these objectives were met by the interventionist. Treatment Fidelity was defined as the percentage of objectives delivered by the interventionist for each wave.
Time Frame: 6-months
Population: Treatment groups of randomized participants in each condition.
Measure: Mean (Standard Deviation); unit: Percentage of unit objectives delivered
Units Other Than Participants: Treatment groups
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 162
Number analyzed (Treatment groups) | 9 | 9
Percentage of unit objectives delivered | 100 (0) | 88.2 (11.0)

47. Secondary Outcome: Habitual Sleep Efficiency
Description: To measure sleep quality we used select questions from the Pittsburgh Sleep Quality Index to calculate habitual sleep efficiency (the percentage of time in bed spent sleeping).
Time Frame: Baseline
Population: Randomized participants who completed the PSQI items
Measure: Median (Inter-Quartile Range); unit: Percentage of time spent in bed sleeping
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 167 | 161
Percentage of time spent in bed sleeping | 87.5 [80.0 to 93.3] | 87.5 [77.8 to 93.3]

48. Secondary Outcome: Habitual Sleep Efficiency
Description: To measure sleep quality we used select questions from the Pittsburgh Sleep Quality Index which allowed the calculation of habitual sleep efficiency (the percentage of time in bed spent sleeping).
Time Frame: 6-months
Population: Randomized participants who completed the PSQI items
Measure: Median (Inter-Quartile Range); unit: Percentage of time spent in bed sleeping
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 128 | 140
Percentage of time spent in bed sleeping | 86.7 [77.8 to 93.9] | 85.7 [80.0 to 93.3]

49. Secondary Outcome: Habitual Sleep Efficiency
Description: as for outcome 48
Time Frame: 12-months
Population: Randomized participants who completed the PSQI items
Measure: Median (Inter-Quartile Range); unit: Percentage of time spent in bed sleeping
Arm/Group | Get Social | Traditional
Number analyzed (Participants) | 116 | 128
Percentage of time spent in bed sleeping | 87.5 [80.0 to 100.0] | 85.7 [77.8 to 89.4]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Get Social | Traditional
All-Cause Mortality (participants affected / at risk) | 0/167 | 0/162
Serious Adverse Events (participants affected / at risk) | 0/167 | 0/162
Other Adverse Events (participants affected / at risk) | 52/167 | 49/162
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Get Social (N=167) | Traditional (N=162)
Musculoskeletal Pain or Injury (Musculoskeletal and connective tissue disorders) | 24 (27) | 24 (25)
Communicable Disease (Cold, Flu, Pneumonia) (General disorders) | 9 (9) | 8 (8)
Procedure/Surgery (Surgical and medical procedures) | 8 (10) | 4 (4)
Cardiac Issue (Cardiac disorders) | 4 (4) | 1 (1)
Gastrointestinal Issue (Gastrointestinal disorders) | 4 (5) | 4 (4)
Diabetes or Blood Glucose Issue (Endocrine disorders) | 3 (3) | 1 (1)
Changed Dose of Antidepressant Medication (Psychiatric disorders) | 1 (1) | 3 (3)
Cancer (General disorders) | 3 (3) | 1 (1)
Gyno/Urological Issue (Renal and urinary disorders) | 2 (2) | 1 (1)
Non-musculoskeletal injury, result of accident (Injury, poisoning and procedural complications) | 2 (2) | 4 (4)
Depression/Anxiety (Psychiatric disorders) | 0 (0) | 2 (2)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0/136 (0) | 2/132 (2) — Assessed in females only
Nerve Condition or Swelling in Legs (General disorders) | 0 (0) | 3 (3)
Eye/Ear Infection (Infections and infestations) | 1 (1) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 1 (1)
Autoimmune Disease (Immune system disorders) | 1 (1) | 0 (0)
Asthma Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Fatty Liver Disease (Hepatobiliary disorders) | 0 (0) | 1 (1)
Bariatric Surgery (Surgical and medical procedures) | 1 (1) | 0 (0)
Lyme Disease (Infections and infestations) | 0 (0) | 1 (1)
Sleep Apnea (General disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-07-24): https://cdn.clinicaltrials.gov/large-docs/18/NCT02646618/Prot_001.pdf
  • Statistical Analysis Plan (2021-02-26): https://cdn.clinicaltrials.gov/large-docs/18/NCT02646618/SAP_002.pdf
  • Informed Consent Form (2018-08-03): https://cdn.clinicaltrials.gov/large-docs/18/NCT02646618/ICF_003.pdf